CLINICAL TRIAL: NCT04832620
Title: Defining Optimal Imaging Strategies for Diagnosis, Treatment, and Treatment Evaluation of Chordomas and Chondrosarcomas of the Axial Skeleton
Brief Title: Image Assisted Optimization of Proton Radiation Therapy in Chordomas and Chondrosarcomas
Acronym: CHIPT
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: HollandPTC (Industry); Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Augustinis D.G. Krol, MD PhD, Radiation oncologist, Leiden University Medical Center
Other Study IDs: 41335
Record Dates: First submitted 2021-03-29; First posted 2021-04-06 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Bone Neoplasm of Vertebral Column; Chordoma; Chondrosarcoma; Magnetic Resonance Imaging; PET-CT; Proton Therapy
Keywords: Chordoma; Chondrosarcoma; MRI; PET-CT; Proton therapy
MeSH Terms: conditions — Chordoma; Chondrosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Chordomas and chondrosarcomas located in the axial skeleton are malignant neoplasms of bone. These tumors share the same clinical challenges, as the effect of the disease is more a function of their local aggressiveness than their tendency to metastasize (20% metastasize). The local aggressive behavior can cause debilitating morbidity and mortality by destruction of nearby located critical neurovascular structures. Imaging has, in addition to histopathology, a role in diagnosis and in guiding (neo)adjuvant and definitive treatment. Despite the low sensitivity to radiotherapy, proton radiotherapy has been successfully used as an adjunct to resection or as definitive treatment for aggressive chordomas and chondrosarcomas, making it a standard indication for proton therapy in the Netherlands.

Chordomas and chondrosarcomas consist, especially after previous therapy, of non-viable and viable tumor components. Identification of these viable components by functional imaging is important to determine the effect of previous therapy, as change in total tumor volume occurs more than 200 days after change of functional imaging parameters.

Objective: The main objective of this study is to determine if functional MRI parameters change within 6 months, and earlier than volumetric changes after start of proton beam therapy. This would allow timely differentiation between affected and unaffected (viable) tumor components, which can be used for therapy adjustment.

Secondary objectives: Determine which set of parameters (PET-CT and secondary MRI) can predict clinical outcome (tumor specific mortality, development of metastases, morbidity secondary to tumor activity and morbidity secondary to treatment); determine what type of imaging can accurately identify viable tumor nodules relative to critical anatomical structures; improving understanding of relevance of changing imaging parameters by correlating these with resected tumor.

Study design: Prospective cohort study Study population: LUMC patients diagnosed with primary or recurrent chordoma or chondrosarcoma in the axial skeleton. A number of 20 new patients per year is expected.

Main study parameters: Volumetric and functional MR imaging parameters including permeability parameters.

Secondary parameters are generated by PET-CT (SUV, MTV and TLG), MR (perfusion, permeability and diffusion), therapy (proton beam dose mapping, surgery) and clinical outcome. End points are disease specific survival, progression free survival (including development of metastases), side effects of treatment, and functional outcome (see CRF). In patients who are treated with surgical resection following neo-adjuvant therapy, the surgical specimen will be correlated with imaging findings.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Treatment and clinical management will not be affected in this study, thus the additional burden, risks, and benefits associated with participation in this study are minimal.

Two extra MRI and one PET-CT examination will be planned during proton therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed with primary or recurrent chordoma or chondrosarcoma in the axial skeleton (clivus, spine and sacrum)
* Accepted for standard proton beam therapy

Exclusion Criteria:

* Diagnosis other than chordoma or chondrosarcoma is made.
* Patient refuses (parts) of the standard treatment protocol.
* Patient refuses MRI due to claustrophobia.
* Patient not suitable for MRI due to the presence of MRI incompatible implants.
* Incapacitated patients.
* Patient doesn't allow coded data to be used for analysis.
* Patient is under 50 years of age.
* Lesion size less than 1cm.
* Patients with WHO 3 and higher.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to HollandPTC, or LUMC, or the Netherlands Committee of Bone tumors, histologically diagnosed with primary or recurrent chordoma or chondrosarcoma in the axial skeleton (clivus, spine and sacrum), and accepted for standard proton beam therapy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Vp(max), Vp(min) | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI permeability parameter - tumor plasma volume

SECONDARY OUTCOMES:
Rel Enhancement (%) | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI perfusion parameter showing the signal enhancement of a pixel of certain dynamic relative to that same pixel in the reference dynamic. The reference dynamic is normally the first, pre-contrast dynamic.
Max Enhancement (%) | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI perfusion parameter showing difference between peak intensity S1 and S0.
Max Rel Enhancement (%) | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI perfusion parameter showing maximum of all relative enhancements over all dynamics
Time of arrival T0 (s) | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI perfusion parameter showing time at which the signal intensity increases for at least 20% compared to the baseline (referred to as initial signal intensity S0).
  The baseline is the average of the signal intensities of all timepoints before the contrast uptake starts.
Time To Peak (s) | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI perfusion parameter showing time till contrast agent bolus reaches peak intensity
Wash In Rate (sˉ¹) | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI perfusion parameter showing maximum slope between T0 and time of peak intensity T1
Wash Out Rate (sˉ¹) | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI perfusion parameter showing maximum slope between time of peak intensity T1 and the end of the measurement
Brevity of Enhancement (s) | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI perfusion parameter showing time between point of maximum wash in rate and maximum wash out rate.
Ktrans | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI permeability parameter - transfer constant between blood plasma and Extravascular Extracellular Space (EES), also called vascular permeability
kep | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI permeability parameter showing rate between EES and blood plasma (also called Tracer Efflux Rate)
Ve | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI permeability parameter showing Extravascular Volume fraction (Leakage space); defined as Ktrans / kep
Area under the curve (AUC) | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI permeability and perfusion parameter showing area Under the Curve of all time curves
mean ADC, Min ADC, Max ADC | At inclusion, 4 and 8 weeks, 5,11,17 and 23 months after the start date of proton therapy treatment
  MRI diffusion parameters
SUV | At inclusion and and 11 months following the start date fo proton therapy
  Standard uptake value extracted from PET-CT imaging
MTV | At inclusion and and 11 months following the start date fo proton therapy
  Metabolic tumor volume extracted from PET-CT imaging
TLG | At inclusion and and 11 months following the start date fo proton therapy
  Total lesion glycolysis extracted from PET-CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Krol, MD PhD, Principal Investigator — LUMC/HollandPTC; Hans Bloem, prof. MD PhD, Principal Investigator — LUMC
Locations (2):
- Netherlands (2):
  - HollandPTC, Delft, South Holland
  - LUMC, Leiden, South Holland